CLINICAL TRIAL: NCT05126758
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Efficacy and Safety of Human Allogeneic Cardiosphere-Derived Cells for the Treatment of Duchenne Muscular Dystrophy
Brief Title: A Study of Deramiocel (CAP-1002) in Ambulatory and Non-Ambulatory Patients With Duchenne Muscular Dystrophy
Acronym: HOPE-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Capricor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAP-1002-DMD-04
Record Dates: First submitted 2021-11-04; First posted 2021-11-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Muscular Dystrophies; Muscular Dystrophy, Duchenne; Muscular Disorders, Atrophic; Muscular Diseases; Neuromuscular Diseases; Genetic Diseases, X-Linked; Genetic Diseases, Inborn; Nervous System Diseases
Keywords: Duchenne Muscular Dystrophy; Cell Therapy; Performance of the Upper Limb; Ambulatory; Non-Ambulatory
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne; Muscular Disorders, Atrophic; Muscular Diseases; Neuromuscular Diseases; Genetic Diseases, X-Linked; Genetic Diseases, Inborn; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Cohort A: placebo-controlled, double-blind, randomized 1:1 (active:placebo); Cohort B: placebo-controlled, double-blind, randomized 1:1 (active:placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Deramiocel (CAP-1002) (Experimental): Cohort A: Approximatetly 29 subjects will receive deramiocel (CAP-1002A) active treatment consisting of 150 million cardiosphere-derived cells (CDCs) via intravenous infusion every 3 months
  Cohort B: Approximately 22 participants will receive deramiocel (CAP-1002B) active treatment consisting of 150 million cardiosphere-derived cells (CDCs) via intravenous infusion every 3 months
  Interventions: Biological: Deramiocel (CAP-1002)
- Placebo (Placebo Comparator): Cohort A: Approximately 29 subjects will receive a Placebo solution via intravenous infusion every 3 months
  Cohort B: Approximately 22 participants will receive a Placebo solution via intravenous infusion every 3 months
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Deramiocel (CAP-1002) — Cohort A: CAP-1002A manufactured in Los Angeles, CA; Cohort B: CAP-1002B manufactured in San Diego, CA
  Other Names: Cardiosphere-Derived Cells (CDCs)
  Arms: Deramiocel (CAP-1002)
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
HOPE-3 is a two cohort, Phase 3, multi-center, randomized, double-blind, placebo-controlled clinical trial evaluating the efficacy and safety of a cell therapy called deramiocel (CAP-1002) in study participants with Duchenne muscular dystrophy (DMD) and impaired skeletal muscle function. Non-ambulatory and ambulatory boys and young men who meet eligibility criteria will be randomly assigned to receive either deramiocel or placebo every 3 months for a total of 4 doses during the first 12 months of the study. All participants will be eligible to receive 4 doses of deramiocel for an additional 12 months as part of an open-label extended assessment period. After completion of the first open-label extension (Months 12-24), subjects who have completed Month 24 are eligible to continue onto a Long-Term Open-Label Extension period that will provide treatment with deramiocel until commercial availability, or until sponsor's decision to terminate the trial, or the participant withdraws consent.

DETAILED DESCRIPTION:
Up to 102 eligible study subjects will participate in this two cohort study. Cohort A will enroll approximately 58 subjects randomized in a 1:1 ratio (active:placebo). Subjects randomized to the active treatment group in Cohort A will receive CAP-1002A (deramiocel manufactured at Capricor's manufacturing facility in Los Angeles, CA). Once Cohort A enrollment is completed, Cohort B enrollment will begin. Cohort B will enroll approximately 44 participants randomized in a 1:1 ratio (active:placebo). Subjects randomized to the active treatment group in Cohort B will receive CAP-1002B (deramiocel manufactured at Capricor's manufacturing facility in San Diego, CA). Both cohorts will include visits at Screening, Baseline/Day 1, Month 1, and Months 3, 6, 9, and 12. Subjects will receive IV infusions of deramiocel or placebo on Day 1 and Months 3, 6, and 9. All subjects will then be eligible to receive additional IV infusions of deramiocel at Month 12, 15, 18, and 21 as part of the open-label phase of the study. All subjects who complete the first open-label extension phase of the study will be eligible to receive additional IV infusions of deramicoel every 3 months in a Long Term Open-Label Extension phase until commercial availability of deramiocel, or until sponsor's decision to terminate the trial, or the participant withdraws consent.

A primary analysis of efficacy and safety will be performed on the double-blind placebo-controlled phase of the study for both Cohort A and Cohort B combined at Month 12 following 4 administrations of deramiocel or placebo.

The primary efficacy endpoint is the mean change from baseline in upper limb function as assessed by Performance of the Upper Limb test, version 2.0 [PUL 2.0] Total Score at the 12-month time point. Secondary endpoints evaluated at the 12-month time point include assessment of changes in cardiac muscle function and structure by cardiac magnetic resonance imaging [cMRI], changes in hand-to-mouth function [eat 10-bites assessed by the Duchenne Video Assessment (DVA)], quality of life assessments, and biomarker analysis for creatine kinase MB isoenzyme (CK-MB).

Safety evaluations will include adverse events, concomitant medications, physical exam, vital signs, and clinical laboratory testing.

An analysis of extended safety and efficacy will be performed in the subsequent open-label phases of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects at least 10 years of age at time of consent who are willing and able to provide informed consent to participate in the trial if ≥ 18 years of age or assent with parental or guardian informed consent if < 18 years of age. If a third-party caregiver is involved, they must provide informed consent.
2. Diagnosis of DMD based on clinical and phenotypic manifestations consistent with DMD (e.g., family history of DMD, elevated creatine kinase, dystrophin muscle biopsy, calf pseudohypertrophy, history of Gowers' sign, and gait impairment before 7 years of age) as confirmed by the Investigator.
3. Confirmatory genetic testing performed to have reached a diagnosis of DMD at any time in the past or currently performed at a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory or equivalent.
4. Performance of the Upper Limb test (PUL) entry item scores 2-6 and total PUL score less than or equal to 40. For Cohort A only: enrollment of patients with PUL entry score 6, Exon 44 skipping amenable, and/or Exon 3 through 7 deletions will be capped at no more than 10% of the total study population (approximately 6 patients with these characteristics).
5. Reduced ability to walk/run (if ambulatory): subjects must take more than 10 seconds for the 10-meter walk/run (i.e., velocity < 1 meter/second).
6. If non-ambulatory, loss of independent ambulation between 10th and 18th year birthday (standing unassisted or ability to take, at most, several steps independently is not considered ambulation). Subjects who are considered non-ambulatory between the ages of 9 and10 may be enrolled with prior approval from the sponsor.
7. Receiving standard of care therapy at an experienced, multidisciplinary DMD center as evidenced by regular cardiac and pulmonary monitoring, systemic glucocorticoid treatment, and at-home range of motion exercises.
8. Treatment with systemic glucocorticoids for at least 12 months and at a stable dose at least 6 months prior to study participation, except for either weight-based dose adjustment or a decrease in steroid dose of ≤ 10% for toxicity. For patients on chronic deflazacort, treatment with an equivalent dose of prednisone or prednisolone for a period of ≤ 30 days to bridge lack of availability of deflazacort during the 6 months prior to randomization is acceptable.
9. Current and up-to-date immunizations according to children and adolescent Centers for Disease Control and Prevention immunization schedule at the discretion of the Investigator.
10. Adequate venous access for parenteral IP infusions and routine blood collection.
11. Assessed by the Investigator as willing and able to comply with the requirements of the trial.
12. Sexually active subjects and their partners who are fertile must agree to use effective method(s) of contraception.

Exclusion Criteria:

1. Left ventricular ejection fraction (LVEF) less than or equal to 35% prior to randomization.
2. Elbow-flexion contractures > 30° in both extremities.
3. Body mass index (BMI) > 45.
4. Percent predicted forced vital capacity (FVC%) < 35% within 6 months prior to randomization.
5. Inability to perform consistent PUL 2.0 measurement within ± 2 points without shoulder domain or within ± 3 points with shoulder domain during paired testing at screening.
6. Risk of near-term respiratory decompensation in the judgment of the Investigator, or the need for initiation of day and night non-invasive ventilator support as defined by serum bicarbonate ≥ 29 mmol/L at screening.
7. History of non DMD-related chronic respiratory disease requiring ongoing or intermittent treatment, including, but not limited to, asthma, bronchitis, and tuberculosis.
8. Acute respiratory illness within 30 days prior to screening and during screening.
9. Initiation of nocturnal non-invasive ventilation within 30 days prior to screening.
10. Planned or anticipated thoracic or spinal surgery within the 6 months following randomization.
11. Planned or anticipated lower extremity surgery within the 6 months following randomization, if ambulatory.
12. Known hypersensitivity to dimethyl sulfoxide (DMSO) or bovine products.
13. Initiation of treatment with metformin or insulin within 3 months prior to randomization.
14. Initiation of treatment with an FDA-approved exon skipping therapy for the treatment of DMD and/or non-weight based adjustments within 12 months prior to randomization.
15. Treatment with human growth hormone within 3 months prior to randomization, unless on a stable dose allowing for weight-based dose adjustments (as determined by the site Investigator) for at least 24 months prior to randomization.
16. Treatment with a cell therapy product within 12 months prior to randomization; any prior exposure to deramiocel will be excluded.
17. Treatment with an investigational product within 6 months prior to randomization.
18. History, or current use, of drugs or alcohol that could impair the ability to comply with participation in the trial.
19. Inability to comply with the investigational plan and follow-up visit schedule for any reason, in the judgment of the investigator.
20. Inability to undergo a cardiac MRI. For Cohort B Only - Subjects with a known hypersensitivity to gadolinium may forgo the LGE assessment but must complete a cardiac MRI without contrast. For Cohort B Only - Subjects who are unable to tolerate gadolinium due to renal insufficiency as measured by an estimated Glomerular Filtration Rate (eGFR) less than 60 mL/min/1.73 m2 may forgo the LGE assessment but must complete a cardiac MRI without contrast.
21. For Cohort B: Subjects with PUL entry score 6, Exon 44 skipping amenable, or Exon 3 through 7 deletions are excluded from participation.

Min Age: 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in the upper limb function | At Month 12
  Mean percent change from baseline in Performance of the Upper Limb test, version 2 (PUL 2.0) Total Score. Items are scored on a three-point scale: 0=unable to perform the item, 1=impaired or performs with compensation, 2=performs task without compensation. Percent change from baseline is calculated as change from baseline divided by baseline score at the subject level.

SECONDARY OUTCOMES:
Change in cardiac muscle function and structure by assessment of left ventricular ejection fraction | At Month 12
  Mean change from baseline in left ventricular ejection fraction as assessed by Cardiac Magnetic Resonance (cMRI) and assessed centrally
Change in mid-level (elbow) upper limb function | At Month 12
  Mean percent change from baseline in mid-level [elbow] upper limb function in Performance of the Upper Limb test, version 2 (PUL 2.0); items are scored on a three-point scale: 0=unable to perform the item, 1=impaired or performs with compensation, 2=performs task without compensation. Percent change from baseline is calculated as change from baseline divided by baseline score at the subject level.
Change in Global Statistical Test (Total GST) combining upper limb function, cardiac muscle function, and patient reported measure of disease severity | At Month 12
  Mean change from baseline in Total GST that combines PUL 2.0 score, LVEF assessment by cMRI, and the Patient Global Impression of Severity (PGI-S)
Change in the number of segments of myocardial scarring (Cohort B only) | at Month 12
  Change in the number of segments of myocardial scarring as observed by late gadolinium enhancement (LGE)
Change in cardiac muscle function and structure by assessment of left ventricular end-systolic volume | At Month 12
  Mean change from baseline in left ventricular indexed end-systolic volume as assessed by Cardiac Magnetic Resonance (cMRI)
Change in cardiac muscle function and structure by assessment of left ventricular ejection fraction in subjects with documented cardiomyopathy | At Month 12
  Mean change from baseline in left ventricular ejection fraction as assessed by Cardiac Magnetic Resonance (cMRI) in subjects with documented cardiomyopathy at baseline.
Change in a global statistical test (Cardiac GST) combining assessments of cardiac muscle function and structure | At Month 12
  Mean change from baseline in Cardiac GST that combines LVEF, LV end-systolic volume index, and LV end-diastolic volume index
Change in percentage of myocardial scarring (Cohort B only) | at Month 12
  Change in percentage of myocardial scarring as observed by late gadolinium enhancement (LGE)
Change in hand-to-mouth function in the context of functional eating | At Month 12
  Mean change from baseline in the functional ability of eating 10 bites evaluated by Duchenne Video Assessment (DVA) using a video record of patient performing the task at home. Physical therapists score the patient's quality of movement in the video using scorecards with pre-specified compensatory movement criteria.
Changes in cardiac inflammation biomarker, creatine kinase MB isoenzyme [CK-MB] | At Month 12
  Mean change from baseline in CK-MB blood levels - MB fraction (% of total CK).

CONTACTS AND LOCATIONS:
Overall Officials: Craig McDonald, MD, Principal Investigator — University of California, Davis; Mark Awadalla, Study Director — Capricor Inc.
Locations (20):
- United States (20):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCSD Altman Clinical and Translational Research Institute, La Jolla, California
  - Children's Hospital of Los Angeles, Division of Neurology, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Missouri Health Care, Columbia, Missouri
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Rare Disease Research NC LLC, Hillsborough, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Health Specialty Care Pavilion, Dallas, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Virginia Children's Hospital, Charlottesville, Virginia
  - Seattle Children's, Seattle, Washington
  - Children's Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No